CLINICAL TRIAL: NCT00830375
Title: Memantine Treatment of Compulsive Buying: An Open-Label Study
Brief Title: Memantine Treatment of Compulsive Buying
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0806M37821
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Results first posted 2012-05-04 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Compulsive Buying
Keywords: Buying; Shopping; Impulse Control
MeSH Terms: conditions — Typhus, Endemic Flea-Borne | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Memantine (Experimental): 10-30mg, memantine
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — 10-30mg, by mouth, daily
  Other Names: Namenda

SUMMARY:
This is an 8-week, open-labe study of memantine in the treatment of compulsive buying.

DETAILED DESCRIPTION:
The goal of the proposed study is to evaluate the efficacy of memantine in the treatment of compulsive buying. Sixteen subjects meeting criteria for compulsive buying will receive 8 weeks of open-label memantine. The hypothesis to be tested is that memantine will be effective and well tolerated in patients with compulsive buying. The proposed study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

ELIGIBILITY:
Inclusion Criteria:

1. men and women age 18-65
2. current CB using the clinician-administered Structured Clinical Interview for Compulsive buying (SCI-CB)
3. buying behavior within 2 weeks prior to enrollment

Exclusion Criteria:

1. infrequent buying (i.e. less than one time per week) that does not meet proposed criteria for CB
2. unstable medical illness or clinically significant abnormalities on laboratory tests or physical examination at screen
3. history of seizures
4. myocardial infarction within 6 months
5. current pregnancy or lactation, or inadequate contraception in women of childbearing potential
6. a need for medication other than memantine with possible psychotropic effects or unfavorable interactions;
7. clinically significant suicidality;
8. current Axis I disorder determined by the SCID and SCID-compatible modules for impulse control disorders, except for nicotine dependence
9. lifetime history of bipolar disorder type I or II, dementia, schizophrenia, or any psychotic disorder determined by SCID
10. current or recent (past 3 months) DSM-IV substance abuse or dependence;
11. positive urine drug screen at screening
12. initiation of psychotherapy or behavior therapy within 3 months prior to study baseline
13. previous treatment with memantine
14. treatment with investigational medication or depot neuroleptics within 3 months, with fluoxetine within 6 weeks, or with other psychotropics within 2 weeks prior to study baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2010-08-01 (Actual); Study Completion 2010-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Grant, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Ambulatory Research Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- See also: Impulse Control Disorders Clinic - University of Minnesota — http://www.impulsecontroldisorders.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: December 2008 - August 2010
Groups:
- Memantine: 10-30mg tablets of memantine taken once daily by mouth
Period: Overall Study
Arm/Group | Memantine
Started | 10
Completed | 9
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Memantine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Yale Brown Obsessive Compulsive Scale Modified for CB (CB-YBOCS)
Description: The CB-YBOCS is a reliable and valid, 10-item, clinician-administered scale that rates buying symptoms within the last seven days, on a severity scale from 0 to 4 for each item (total scores range from 0 to 40 with higher scores reflecting greater illness severity). Scores ranging from 0 to 10 reflect minimal or mild symptoms; scores from 11 to 20 suggest moderate symptoms; severe symptoms are associated with scores from 21 to 30; and scores greater than 30 reflect extreme buying symptoms
Time Frame: from study start to study end (8-weeks) and is Investigator rated
Population: Reported scores are Mean and standard deviation for Subjects last visit (Week 8 or last-observation carried forward).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 10
units on a scale | 22 (4)

ADVERSE EVENTS:
Arm/Group | Memantine
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No